CLINICAL TRIAL: NCT04340778
Title: Comparative Safety and Efficacy of Vaginal Dinoprostone Versus Lidocaine-prilocaine Cream in Copper IUD Insertion in Nulliparous Women: a Randomized Controlled Trial
Brief Title: Comparative Safety and Efficacy of Vaginal Dinoprostone Versus Lidocaine-prilocaine Cream in Copper IUD Insertion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dinoprostone vs LP cream
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Contraception

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vaginal dinoprostone (Experimental): vaginal dinoprostone 3 mg will be given 3 hours before copper IUD insertion plus inert placebo cream will be applied on the cervix at the time of IUD insertion.
  Interventions: Drug: vaginal dinoprostone
- lidocaine prilocaine cream (Active Comparator): Lidocaine-prilocaine Cream will be applied on the cervix at the time of copper IUD insertion plus vaginal placebo tablet 3 hours before IUD insertion
  Interventions: Drug: Lidocaine-prilocaine Cream
- placebo (Placebo Comparator): inert placebo Cream will be applied on the cervix at the time of copper IUD insertion plus vaginal placebo tablet 3 hours before IUD insertion
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: vaginal dinoprostone — vaginal dinoprostone 3 mg will be given 3 hours before copper IUD insertion plus inert placebo cream will be applied on the cervix at the time of IUD insertion
  Arms: vaginal dinoprostone
Drug: Lidocaine-prilocaine Cream — Lidocaine-prilocaine Cream will be applied on the cervix at the time of IUD insertion plus vaginal placebo tablet will be given 3 hours prior to IUD insertion
  Arms: lidocaine prilocaine cream
Drug: placebo — inert placebo Cream will be applied on the cervix at the time of IUD insertion plus vaginal placebo tablet will be given 3 hours prior to IUD insertion
  Arms: placebo

SUMMARY:
the aim of the present study is to Compare Safety and Efficacy of Vaginal dinoprostone Versus Lidocaine-prilocaine Cream in copper IUD Insertion in nulliparous women: a randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women requesting copper IUD insertion

Exclusion Criteria:

* multiparous women, active vaginal or cervical infections and contraindications to IUD Insertion.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2020-04-30 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-09-05 (Estimated)

PRIMARY OUTCOMES:
pain during IUD insertion: visual analog scale | 5 minutes
  pain during copper IUD insertion evaluated by 10 cm visual analog scale where 0 denotes no pain and 10 cm denotes the worst pain imaginable

SECONDARY OUTCOMES:
duration of insertion | 5 minutes
  duration of insertion from speculum in to speculum out